CLINICAL TRIAL: NCT01677091
Title: Effectiveness of a Balance Rehabilitation Program With Sensory Recalibration After Stroke: A Randomized Controlled Trial.
Brief Title: Balance Rehabilitation With Sensory Recalibration After Stroke
Acronym: AVCPOSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-A00667-36
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Left-sided Hemiplegia Affecting Dominant Side as Late Effect of Cerebrovascular Accident
Keywords: Balance,Hemiplegia,Cervical vibration,Prism adaptation,Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control group (Active Comparator): This group will benefit from conventional rehabilitation
  Interventions: Other: Conventional rehabilitation
- Cervical vibration (Experimental): This group will benefit from a daily 20 minutes session, with vibration of neck muscles during 10 minutes
  Interventions: Other: Cervical vibration
- Prism adaptation (Experimental): This group will benefit from a daily 20 minutes session, with prism adaptation during 10 minutes
  Interventions: Other: Prism adaptation
- Cervical vibration + Prism adaptation (Experimental): This group will receive a daily 30 minutes session, with cervical vibration during 10 minutes + prism adaptation during 10 minutes
  Interventions: Other: Cervical vibration; Other: Prism adaptation

INTERVENTIONS:
Other: Cervical vibration — Vibration of neck muscles during 10 minutes
  Arms: Cervical vibration; Cervical vibration + Prism adaptation
Other: Prism adaptation — Prism adaptation during 10 minutes
  Arms: Cervical vibration + Prism adaptation; Prism adaptation
Other: Conventional rehabilitation — conventional rehabilitation
  Arms: Control group

SUMMARY:
The main objective of this study is to test the effectiveness of a rehabilitation program with cervical vibration and/or prism adaptation in patients with left hemiplegia on balance.

DETAILED DESCRIPTION:
Imbalance is particularly severe after a Cerebral Vascular Accident because they not only limit the capacity of transfer and are a source of falls but also represent an obstacle to the acquisition of autonomy.

When the brain lesion is located in the right hemisphere, the prognosis in terms of equilibrium is worse probably because of the presence of disorders of spatial cognition. These disorders of spatial cognition are manifested by a distortion of the mental representation of space and body in space that probably cause a deviation of the position of the center of pression on platform. This component of balance disorders secondary to disruption of spatial cognition, do not benefit at present from specific rehabilitative treatment despite the severity of the consequences.

But the application of sensory manipulations has proven its effectiveness on visuospatial neglect that is another disorder of spatial cognition closed to the pathophysiology of balance disorders after right brain lesion. Sensory manipulations decrease the distortion of internal representations of the body in space by restoring the symmetry of sensory inputs. Some of these manipulations (visual manipulation by wearing prisms and proprioceptive manipulations) are also effective on the immediate correction of postural imbalances on force platform and disorders of spatial perception.

We therefore believe that the approach by repeated sensory manipulation is a new promising way of research for the rehabilitative treatment of balance disorders secondary to disorders of spatial cognition. As the mechanisms of action and the structures involved during proprioceptive vibration of neck muscles and during visual prism adaptation are different, we believe that the combination of these two types of sensory manipulations will permit to obtain a greater and longer lasting effect than a lonely manipulation. The concomitant evaluation of the bias on postural platform and the perception of the body axis will allow us to assess the impact of such rehabilitation on the disorders of spatial representation and so better understand the mechanisms of action of sensory manipulations.

The main objective of this study is to test the effectiveness of a rehabilitation program with cervical vibration (V) and / or prism adaptation (P) in patients with left hemiplegia on balance at the end of the intervention (day14).

Secondary objectives are to test:

* The immediate effect (day 0) on force platform evaluation of balance,
* Maintaining the gain at 3 months and 6 months on balance,
* Effectiveness at day 14 on negligence
* Maintaining the gain at 3 months and 6 months on neglect,
* Effectiveness at day 14 on functional abilities,
* Maintaining the gain at 3 months and 6 months on functional abilities,
* Understanding the mechanisms of action of each of the sensory manipulations by assessing changes in perceptions of space, after rehabilitation programs (day 14) and at 3 months and 6 months.
* To evaluate the evolution of motility, sensitivity and spasticity in the various assessments.

During the 15 days rehabilitation performed for the study, the upper and lower limbs motor rehabilitation will last less than one hour and a half, and will exclude instrumental techniques of balance rehabilitation, sensory manipulations, virtual reality, strain-induced therapy.

Moreover, an ancillary study will be performed to study the immediate neurofunctional effect of vibratory stimulation, in right brain-damaged patients with imbalance and in healthy volunteers, through the assessment of cerebral activation changes in MRI. The secondary objectives of this ancillary study are to test the neurofunctional effect of repeated vibratory stimulation in right brain-damaged patients, describe the relationship between cerebral activation changes and evolution of balance, and describe the areas of the brain activated by vibratory stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Right unilateral supratentorial ischemic or hemorrhagic lesion
* Adult (age ≥ 18 years) under 80 years
* Stroke

  * older than 9 months
  * with or without hemianopsia
  * with or without visuospatial hemineglect
* The first symptomatic episode
* Standing balance ≥ 30 sec unaided
* Percentage of weight rests on the hemiplegic lower limb below 40% of body weight (on a platform of strength)
* Written informed consent of the patient or a member of his entourage (in the case of patients with motor difficulties)

Exclusion Criteria:

* Orthopedic, rheumatologic or visual disorders affecting the distribution of the center of pressure while standing
* Visual disorder that does not allow assessment of the longitudinal axis or visual straight ahead
* Ischemic or hemorrhagic brain stem lesion
* Trouble for understanding protocol procedures

Inclusion Criteria for the healthy volunteers (ancillary study) :

* Age ≥ 18 years, right-handed, sex and age-matched (+/- 5 years) to the patients of the coordinating center
* Able to get an MRI
* With no imbalance
* With no visual disorder impacting the repartition of the center of pression when standing up, or that does not allow assessment of the longitudinal axis or visual straight ahead
* Written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-05-05 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the deviation of the mean position of center of pressure (CP) (eyes closed) on the mediolateral axis (mm) assessed by posturography after intervention. | Day 14

SECONDARY OUTCOMES:
Evaluation of balance | Day 0, Day 14, Month 3, Month 6
  * Postural Assessment Scale for Stroke
  * Scale for Contraversive Pushing
  * Berg Balance Scale
  * Timed Up and Go
  * Measurement performed on the platform of strength:
    * surface of the center of mass displacement
    * deviation of the mean position of the center pressure on the anteroposterior axis
    * standard deviation of the average displacement of the center pressure on the mediolateral axis and the anteroposterior axis,
    * percentage of support on the hemiplegic lower limb.
Evaluation of functional capacity | Day 0, Day 14, Month 3, Month 6
  * Barthel Index (Day 0, Day 14, Month 3, Month 6)
  * Number of hours of help at home (Month 3, Month 6)
  * Total Duration of hospitalization since the Cerebral Vascular Accident (Month 3, Month 6)
Evaluation of negligence | Day 0, Day 14, Month 3, Month 6
  * Bell test,
  * Bisection test,
  * Scale of Catherine Bergego,
  * OTA test
  * Test of bodily neglect.
Understanding the mechanisms of sensory manipulations | Day 0, Day 14, Month 3, Month 6
  * Evaluation of longitudinal axis by a fluorescent bar movement in front of the patient through a computerized system.
  * Haptic Straight Ahead using a graduated table on which the subject moves his hand blindfolded.

OTHER OUTCOMES:
Time since stroke | day 0
Extent of the injury and localization of brain injury | >2 months after hemiplegia
  Assessed by morphological MRI with DT1, TSE T2 and flair sequences, to achieve a morphological analysis of the lesion. The MRI will be read back by Rennes.
Severity of hemiplegia | day 0
  motility index, Barthel
Study the effect of vibratory stimulation by studying changes in brain activity in particular areas of interest involved in the representation of the body (ancillary study) | Day 0, Week 3
  Day 0 : Functional MRI analysis for the patients included in the coordinating center (Rennes).
  Week 3 : Among these patients, a second functional MRI will be performed for the first 10 patients of the cervical vibration group and first 10 patients of the conventional rehabilitation group, and for 20 age and sex-matched healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle BONAN, PU PH, Principal Investigator — Rennes University Hospital
Locations (8):
- France (8):
  - CHU Grenoble, Grenoble
  - CHU Lille, Lille
  - CHU Lyon, Lyon
  - IRF Nancy, Nancy
  - CHU Lariboisière-Saint Louis Paris, Paris
  - Centre de Rééducation de Kerpape, Ploemeur
  - CHU Reims, Reims
  - CHU Rennes-Pontchaillou, Rennes

REFERENCES:
- [Result] Leplaideur S, Moulinet-Raillon A, Duche Q, Chochina L, Jamal K, Ferre JC, Bannier E, Bonan I. The Neural Bases of Egocentric Spatial Representation for Extracorporeal and Corporeal Tasks: An fMRI Study. Brain Sci. 2021 Jul 22;11(8):963. doi: 10.3390/brainsci11080963. PMID 34439582
- [Result] Jamal K, Leplaideur S, Rousseau C, Cordillet S, Raillon AM, Butet S, Cretual A, Bonan I. The effects of repetitive neck-muscle vibration on postural disturbances after a chronic stroke. Neurophysiol Clin. 2020 Sep;50(4):269-278. doi: 10.1016/j.neucli.2020.01.005. Epub 2020 Mar 31. PMID 32245547
- [Derived] Leplaideur S, Allart E, Chochina L, Perennou D, Rode G, Boyer FC, Paysant J, Yelnik A, Jamal K, Duche Q, Morcet JF, Laviolle B, Combes B, Bannier E, Bonan I. Neck muscle vibration and prism adaptation fail to improve balance disturbances after stroke: A multicentre randomised controlled study. Ann Phys Rehabil Med. 2024 Oct;67(7):101871. doi: 10.1016/j.rehab.2024.101871. Epub 2024 Aug 21. PMID 39173550